CLINICAL TRIAL: NCT01321125
Title: Comparative Study of 2% Chlorhexidine Gluconate in 70% Isopropyl Alcohol Against 10% Sodium Hypochlorite as Skin Antiseptics in Human Volunteers
Brief Title: Chlorhexidine Against Sodium Hypochlorite as Skin Antiseptics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Antisepsia Central (Industry)
Responsible Party: Principal Investigator, Alejandro E. Macias, MD, Universidad de Guanajuato
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2011UGTO372
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2011-09

CONDITIONS: Infectious Diseases
Keywords: Antiseptics; Administration cutaneously; Chlorine compounds; Anti-infecting agents, local
MeSH Terms: conditions — Communicable Diseases | interventions — chlorhexidine gluconate; 2-Propanol; Hypochlorous Acid; Povidone-Iodine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole group of 30 volunteers (Experimental): The arm is composed of 30 human volunteers to test 2% chlorhexidine gluconate in 70% isopropyl alcohol (ChloraPrep ®, Enturia, Texas, USA ), hypochlorite 10% of electrochemical production (Except 10% ®, Pisa, Guadalajara, Mexico), and two controls.
  Interventions: Biological: Bacterial culture of the prepared skin's areas; Other: Preparing skin's areas to be tested
- test group of substantivity (Experimental): The arm is composed of 10 human volunteers to test 2% chlorhexidine gluconate in 70% isopropyl alcohol (ChloraPrep ®, Enturia, Texas, USA ), hypochlorite 10% of electrochemical production (Except 10% ®, Pisa, Guadalajara, Mexico), and 10% povidone-iodine (Isodine Solucion ®, Boehringer-Ingelheim Promeco, Mexico City)
  Interventions: Biological: Antiseptic substantivity

INTERVENTIONS:
Biological: Bacterial culture of the prepared skin's areas — Cultures were taken with a scrub-cup of 5cm2 of internal area pressed over the skin previously prepared, then it was added a 3mL of culture broth (C/E neutralizing broth (D/E Neutralizing Broth, DIFCO TM) containing a neutralizing agent and a detergent agent (1% solution tween-80) as washing solution. The skin was scrub with a sterile rubber policeman for 2 minutes, and the procedure was conducted once again. Both aliquots were gathered together in a sterile tube, and a sample of 50mL was spread in a plate containing a neutralizing agar (D/E neutralizing Agar, DIFCO TM) and incubated at 35°C for 72 hrs. After incubation, the colonies were counted.
  Other Names: Neutralizing agar; Neutralizing broth
  Arms: Whole group of 30 volunteers
Other: Preparing skin's areas to be tested — Two antiseptics (2% chlorhexidine gluconate in 70% isopropyl alcohol and 10% sodium hypochlorite) and two controls were tested as skin antiseptics. The intervention consisted of preparing four skin's areas with the antiseptic or the control, two in each arm of the volunteer. These ones were approximately 25cm2 on the forearm for each antiseptic or control. The antiseptic or control were applied in an outward circular motion using a swab that was soaked with the solution. The solution was kept on the skin for 60 seconds before the bacterial culture was conducted. Every volunteer were studied in three separate occasions, alternating the four areas in every subsequent test, so every area was studied with each control or antiseptic.
  Other Names: Chloraprep (R); Except (R)
  Arms: Whole group of 30 volunteers
Biological: Antiseptic substantivity — Three antiseptics will be tested: 2% chlorhexidine gluconate in 70% isopropyl alcohol, 10% sodium hypochlorite and 10% povidone-iodine, each one will be applied on the surface of one fingertip each, and will be allow to dry for 60 seconds, then the remaining antiseptic on the skin will be wash out with distilled water. The evaluated zones will be dried with sterile gauze, and then will be covered with sterile gauze for two hours. After this period, each finger will be placed for 30 seconds on an agar plate, which will be inoculated whit an ATCC E. coli. The plate will be incubated at 35ºC for 72 hrs. After incubation, a blinded technician will report the presence or absence of bacterial growth
  Other Names: 2% chlorhexidine gluconate in 70% isopropyl alcohol (ChloraPrep ®, Enturia, Texas, USA ); hypochlorite 10% of electrochemical production (Except 10% ®, Pisa, Guadalajara, Mexico); 10% povidone-iodine (Isodine Solucion ®, Boehringer-Ingelheim Promeco, Mexico City); Muller Hinton agar plate (BD/BBL ™, México City, México).
  Arms: test group of substantivity

SUMMARY:
The physicians have few options for skin antisepsis. Alternatives for common use antiseptics are costly or ineffective. In order to have more options, this study is needed. The investigators want to know if there are differences between the use of 2% chlorhexidine gluconate in 70% isopropyl alcohol or 10% sodium hypochlorite.

DETAILED DESCRIPTION:
Sodium hypochlorite at 10% has been widely used as antiseptic in patients on dialysis as well as for irrigation of wounds and burns. Since it has been used successfully in caring for the exit side of hemodialysis catheters, it is reasonable to propose its use for the insertion and care of central intravascular catheters, as well as for skin preparation before surgery. Alternatives for povidone-iodine, which is the agent most commonly used, are costly or ineffective. In a recent study perform by our group it was demonstrated that 10% sodium hypochlorite was not inferior than povidone-iodine.

It has been demonstrated as well that 2% chlorhexidine gluconate in 70% isopropyl alcohol is superior to povidone-iodine. The aim of this study is to know if 10% sodium hypochlorite has a similar effect that the best current option for skin antisepsis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers

Exclusion Criteria:

* History of skin allergies or atopy, as well as reactions to soaps, chlorine or latex

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the efficacy of 2% chlorhexidine gluconate in 70% isopropyl alcohol and 10% sodium hypochlorite | 24 hours
  Compare decrease in colony forming units in cultures of samples taken with both antiseptics

SECONDARY OUTCOMES:
Presence of skin reactions for the 2% chlorhexidine gluconate in 70% isopropyl alcohol | 24 hours
  Presence of allergy or any reaction at 24 hours after the antiseptic application.
Presence of allergy or any reaction at 24 hours after the antiseptic application. | 24 hours
  Presence of allergy or any reaction at 24 hours after the antiseptic application.
Bacterial count of skin cultures for the 2% chlorhexidine gluconate in 70% isopropyl alcohol | 24 hours
  Bacterial colony count of skin cultures to determine antiseptic properties. After incubation, a blinded technician will count the colonies to determine the colony-forming units per square centimeter (CFU/cm2) of skin.
Bacterial count of skin cultures for the 10% sodium hypochlorite | 24 hours
  Bacterial colony count of skin cultures to determine antiseptic properties. After incubation, a blinded technician will count the colonies to determine the colony-forming units per square centimeter (CFU/cm2) of skin.
Bacterial count of skin cultures for the control 1 | 24 hours
  Scrub with saline solution. Bacterial colony count of skin cultures to determine antiseptic properties. After incubation, a blinded technician will count the colonies to determine the colony-forming units per square centimeter (CFU/cm2) of skin.
Bacterial count of skin cultures for the control 2 | 24 hours
  Sample taken without wash. Bacterial colony count of skin cultures to determine antiseptic properties. After incubation, a blinded technician will count the colonies to determine the colony-forming units per square centimeter (CFU/cm2) of skin.
Evaluation of antiseptic substantivity | 24 hours
  Explore the extended antiseptic activity provide by 2% chlorhexidine gluconate in 70% isopropyl alcohol, 10% sodium hypochlorite and 10% povidone-iodine, by evaluating bacterial grow inhibition in an agar plate.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro E Macias, M. D., Principal Investigator — Universidad de Guanajuato
Locations (1):
- University of Guanajuato School of Medicine, León, Guanajuato, Mexico